CLINICAL TRIAL: NCT07212608
Title: Wearable Gait Interventions for Augmenting Paretic Propulsion: Towards Personalized Post-Stroke Gait Rehabilitation
Brief Title: Personalized Post-Stroke Gait Rehabilitation Interventions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University Charles River Campus (Other)
Collaborators: Harvard University (Other); American Heart Association (Other); National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH)
Responsible Party: Principal Investigator, Lou Awad, PT, DPT, PhD, Assistant Professor, Boston University Charles River Campus
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 5715-FEX; U54EB015408 (NIH); 830019 (Other Grant/Funding Number: American Heart Association Pre-Doctoral Fellowship)
Record Dates: First submitted 2025-03-28; First posted 2025-10-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Stroke
Keywords: Exosuit; Neuroprosthesis; Soft Robotics; Wearable Robots; Gait Rehabilitation; Propulsion; Functional Electrical Stimulation (FES); Stroke; Neuromuscular Control
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: All participants will complete a baseline evaluation followed by two training days in a randomly assigned order. The training days are randomized between i) propulsion neuroprosthesis, ii) soft robotic exosuit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Exosuit Training (Experimental): A single 30-minute training of goal-directed overground walking practice at a moderately fast speed with a soft robotic exosuit powered on and off. Shorter overground and treadmill evaluations without the exosuit will be completed immediately before and after the training.
  Interventions: Device: Soft robotic exosuit
- Neuroprosthesis Training (Active Comparator): A single 30-minute training of goal-directed overground walking practice at a moderately fast speed with the propulsion neuroprosthesis powered on and off. Shorter overground and treadmill evaluations without neurostimulation will be completed immediately before and after the training.
  Interventions: Device: Propulsion neuroprosthesis

INTERVENTIONS:
Device: Soft robotic exosuit — A soft robotic exosuit is a textile-based system worn on the waist and paretic lower limb that provides assistive torques via cables connecting the front and back of the ankle to anchor points on the shank. The exosuit provides dorsiflexion assistance during swing phase for foot clearance and plantarflexion assistance during stance phase for propulsion delivered synchronously based on integrated sensors detecting the wearer's gait pattern.
  Arms: Exosuit Training
Device: Propulsion neuroprosthesis — A neuroprosthesis is a textile-based, surface electrical stimulation system worn on the waist and paretic lower limb that delivers stimulation assistance via electroconductive pads placed on the skin over the target muscles. The neuroprosthesis provides coordinated dorsiflexor stimulation during swing phase for foot clearance and plantarflexor stimulation during stance phase for propulsion, delivered synchronously based on integrated sensors detecting the wearer's gait pattern.
  Arms: Neuroprosthesis Training

SUMMARY:
The objective of this study is to understand whether certain post-stroke patient subsets, identified from clinical, biomechanical, and neuromuscular characteristics, preferentially respond to different walking rehabilitation interventions that augment paretic limb propulsion (e.g., soft robotic exosuits or electrical stimulation neuroprostheses). The results of this work could improve post-stroke gait recovery outcomes by informing clinical decision-making to better match patients with rehabilitation devices tailored to their specific gait characteristics.

DETAILED DESCRIPTION:
Stroke is a leading cause of long-term disability that results in slow, asymmetrical, and inefficient walking. Personalized treatments matching patients to the treatments with which they are most likely to respond are not typical but are necessary to maximize recovery.

Post-stroke hemiparesis is commonly associated with reduced paretic limb propulsion that leads to slower, less efficient walking patterns. Our team has developed and tested two rehabilitation technologies targeting paretic propulsion: i) a soft robotic exosuit that uses cables to mechanically assist ankle dorsiflexion and plantarflexion during walking; ii) a neuroprosthesis that uses functional electrical stimulation (FES) to activate the dorsiflexor and plantarflexor muscles during walking. Both technologies aim to safely improve walking speed and paretic propulsion. The objective of this study is to evaluate if certain post-stroke patient subsets, identified from baseline clinical, biomechanical, and neuromuscular characteristics, preferentially respond to propulsion rehabilitation using soft robotic exosuits or electrical stimulation neuroprostheses.

Twenty participants with chronic (>6 months) stroke will complete one baseline gait evaluation in the laboratory and two gait training sessions: i) an exosuit day and ii) a neuroprosthesis day. Each visit will include walking with/without the respective technology.

The primary aim of this study is to identify predictors of a therapeutic response (i.e., improvement in walking speed) to determine whether certain patient subsets preferentially respond to the exosuit or the neuroprosthesis. We will evaluate baseline clinical, biomechanical, and neuromuscular abilities as potential predictors of a response. We hypothesize that a subset of individuals will respond preferentially to each intervention and that baseline measures of gait function will predict responders to each intervention.

A secondary aim of this study is to determine the rehabilitation mechanism underlying improved walking speed after walking with the propulsion exosuit and the neuroprosthesis. Improvements in walking speed can be achieved through recovery (e.g., increased propulsion symmetry) or compensation (e.g., increased nonparetic propulsion). We will independently evaluate the underlying biomechanical changes contributing to improvements in speed and metabolic cost. We hypothesize that both the exosuit and neuroprosthesis will promote improved speed via recovery of paretic propulsion.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a stroke event occurring at least 6 months ago
* Observable gait deficits
* Independent ambulation for at least 30 meters (using an assistive device as needed but without a rigid brace or ankle foot orthosis)
* Passive ankle dorsiflexion range of motion to neutral with the knee extended
* Ability to follow a 3-step command
* Resting heart rate between 40-100 bpm
* Resting blood pressure between 90/60 and 170/90 mmHg
* NIH Stroke Scale Question 1b score > 1 and Question 1c score > 0
* HIPAA authorization to allow communication with healthcare provider
* Medical clearance by a physician

Exclusion Criteria:

* Severe aphasia or inability to communicate with investigators
* Neglect or hemianopia
* Score of >1 on question 1b and >0 on question 1c on the NIH Stroke Scale
* Serious comorbidities that may interfere with ability to participate in the research (e.g., musculoskeletal, cardiovascular, pulmonary)
* Pacemakers or similar electrical implants that could be affected by the FES
* Pressure ulcers or skin wounds located near human-device interface sites
* More than 2 unexplained falls in the previous month
* Actively receiving physical therapy for walking

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2022-09-13 (Actual); Primary Completion 2025-04-24 (Actual); Study Completion 2025-04-24 (Actual)

PRIMARY OUTCOMES:
Unassisted Overground Comfortable Walking Speed (Exosuit Day) | Periprocedural (Before); Periprocedural (After)
  Walking speed without assistance measured at a self-selected comfortable pace using the 10-Meter Walk Test on the training day with the soft robotic exosuit.
Unassisted Overground Fast Walking Speed (Exosuit Day) | Periprocedural (Before); Periprocedural (After)
  Walking speed without assistance measured at a self-selected fast pace using the 10-Meter Walk Test on the training day with the soft robotic exosuit.
Unassisted Paretic Propulsion on Treadmill (Exosuit Day) | Periprocedural (Before); Periprocedural (After)
  Paretic propulsion during walking on the treadmill without assistance on the training day with the soft robotic exosuit at a speed determined by the average walking speed during the 6-Minute Walk Test on the Baseline Evaluation. Paretic propulsion was calculated as the peak anterior-posterior ground reaction force of the paretic limb.
Unassisted Energy Efficiency on Treadmill (Exosuit Day) | Periprocedural (Before); Periprocedural (After)
  Energy efficiency during walking on the treadmill without assistance on the training day with the soft robotic exosuit at a speed determined by the average walking speed during the 6-Minute Walk Test on the Baseline Evaluation. Energy efficiency is measured using indirect calorimetry on a breath-by-breath basis and is calculated as the negative net energy cost of walking with respect to standing rest.
Unassisted Overground Comfortable Walking Speed (Neuroprosthesis Day) | Periprocedural (Before); Periprocedural (After)
  Walking speed without assistance measured at a self-selected comfortable pace using the 10-Meter Walk Test on the training day with the propulsion neuroprosthesis.
Unassisted Overground Fast Walking Speed (Neuroprosthesis Day) | Periprocedural (Before); Periprocedural (After)
  Walking speed without assistance measured at a self-selected fast pace using the 10-Meter Walk Test on the training day with the propulsion neuroprosthesis.
Unassisted Paretic Propulsion on Treadmill (Neuroprosthesis Day) | Periprocedural (Before); Periprocedural (After)
  Paretic propulsion during walking on the treadmill without assistance on the training day with the propulsion neuroprosthesis at a speed determined by the average walking speed during the 6-Minute Walk Test on the Baseline Evaluation. Paretic propulsion was calculated as the peak anterior-posterior ground reaction force of the paretic limb.
Unassisted Energy Efficiency on Treadmill (Neuroprosthesis Day) | Periprocedural (Before); Periprocedural (After)
  Energy efficiency during walking on the treadmill without assistance on the training day with the propulsion neuroprosthesis at a speed determined by the average walking speed during the 6-Minute Walk Test on the Baseline Evaluation. Energy efficiency is measured using indirect calorimetry on a breath-by-breath basis and is calculated as the negative net energy cost of walking with respect to standing rest.

SECONDARY OUTCOMES:
Unassisted Overground Paretic Propulsion at Comfortable Speed (Exosuit Day) | Periprocedural (Before); Periprocedural (After)
  Paretic propulsion during walking without assistance at a self-selected comfortable pace during the 10-Meter Walk Test on the training day with the soft robotic exosuit. Paretic propulsion was calculated as the peak anterior-posterior ground reaction force of the paretic limb.
Unassisted Overground Paretic Trailing Limb Angle at Comfortable Speed (Exosuit Day) | Periprocedural (Before); Periprocedural (After)
  Paretic trailing limb angle during walking without assistance at a self-selected comfortable pace during the 10-Meter Walk Test on the training day with the soft robotic exosuit. Paretic trailing limb angle is the peak angle that the paretic limb makes during terminal stance phase with respect to vertical. Trailing limb angle is measured from the fifth metatarsal head to the greater trochanter with respect to vertical.
Unassisted Overground Paretic Propulsion at Fast Speed (Exosuit Day) | Periprocedural (Before); Periprocedural (After)
  Paretic propulsion during walking without assistance at a self-selected fast pace during the 10-Meter Walk Test on the training day with the soft robotic exosuit. Paretic propulsion was calculated as the peak anterior-posterior ground reaction force of the paretic limb.
Unassisted Overground Paretic Trailing Limb Angle at Fast Speed (Exosuit Day) | Periprocedural (Before); Periprocedural (After)
  Paretic trailing limb angle during walking without assistance at a self-selected fast pace during the 10-Meter Walk Test on the training day with the soft robotic exosuit. Paretic trailing limb angle is the peak angle that the paretic limb makes during terminal stance phase with respect to vertical. Trailing limb angle is measured from the fifth metatarsal head to the greater trochanter with respect to vertical.
Unassisted Paretic Trailing Limb Angle on Treadmill (Exosuit Day) | Periprocedural (Before); Periprocedural (After)
  Paretic trailing limb angle during walking on the treadmill without assistance on the training day with the soft robotic exosuit at a speed determined by the average walking speed during the 6-Minute Walk Test on the Baseline Evaluation. Paretic trailing limb angle is the peak angle that the paretic limb makes during terminal stance phase with respect to vertical. Trailing limb angle is measured from the fifth metatarsal head to the greater trochanter with respect to vertical.
Unassisted Overground Paretic Propulsion at Comfortable Speed (Neuroprosthesis Day) | Periprocedural (Before); Periprocedural (After)
  Paretic propulsion during walking without assistance at a self-selected comfortable pace during the 10-Meter Walk Test on the training day with the propulsion neuroprosthesis. Paretic propulsion was calculated as the peak anterior-posterior ground reaction force of the paretic limb.
Unassisted Overground Paretic Trailing Limb Angle at Comfortable Speed (Neuroprosthesis Day) | Periprocedural (Before); Periprocedural (After)
  Paretic trailing limb angle during walking without assistance at a self-selected comfortable pace during the 10-Meter Walk Test on the training day with the propulsion neuroprosthesis. Paretic trailing limb angle is the peak angle that the paretic limb makes during terminal stance phase with respect to vertical. Trailing limb angle is measured from the fifth metatarsal head to the greater trochanter with respect to vertical.
Unassisted Overground Paretic Propulsion at Fast Speed (Neuroprosthesis Day) | Periprocedural (Before); Periprocedural (After)
  Paretic propulsion during walking without assistance at a self-selected fast pace during the 10-Meter Walk Test on the training day with the propulsion neuroprosthesis. Paretic propulsion was calculated as the peak anterior-posterior ground reaction force of the paretic limb.
Unassisted Overground Paretic Trailing Limb Angle at Fast Speed (Neuroprosthesis Day) | Periprocedural (Before); Periprocedural (After)
  Paretic trailing limb angle during walking without assistance at a self-selected fast pace during the 10-Meter Walk Test on the training day with the propulsion neuroprosthesis. Paretic trailing limb angle is the peak angle that the paretic limb makes during terminal stance phase with respect to vertical. Trailing limb angle is measured from the fifth metatarsal head to the greater trochanter with respect to vertical.
Unassisted Paretic Trailing Limb Angle on Treadmill (Neuroprosthesis Day) | Periprocedural (Before); Periprocedural (After)
  Paretic trailing limb angle during walking on the treadmill without assistance on the training day with the propulsion neuroprosthesis at a speed determined by the average walking speed during the 6-Minute Walk Test on the Baseline Evaluation. Paretic trailing limb angle is the peak angle that the paretic limb makes during terminal stance phase with respect to vertical. Trailing limb angle is measured from the fifth metatarsal head to the greater trochanter with respect to vertical.

OTHER OUTCOMES:
Stroke Chronicity | Baseline (Day 1)
  Length of time since onset of stroke.
Six-Minute Walk Test Distance | Baseline (Day 1)
  Distance walked during the Six-Minute Walk Test (6MWT), a clinical assessment measuring walking endurance.
Fugl-Meyer Assessment of Motor Recovery After Stroke | Baseline (Day 1)
  Score on the Fugl-Meyer Assessment - Lower Extremity (FMA-LE). The FMA-LE includes a series of short activities that are assessed by a physical therapist to evaluate post-stroke recovery.
Plantarflexor Central Drive | Baseline (Day 1)
  Plantarflexor central drive captures the percentage of the plantarflexor muscle's total force-generating capacity that can be voluntarily controlled by an individual with a neurological injury. Central drive is calculated as the ratio of the maximum voluntary isometric contraction (MVIC) to the maximum force generating ability (MFGA).

CONTACTS AND LOCATIONS:
Overall Officials: Louis N Awad, PT, PhD, Principal Investigator — Boston University
Locations (1):
- Boston University Neuromotor Recovery Laboratory, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Awad LN, Bae J, O'Donnell K, et al. Soft exosuits increase walking speed and distance after stroke. In: International Symposium on Wearable Robotics and Rehabilitation (WeRob). Houston, TX: IEEE; 2; 2017.
- [Background] Awad LN, Bae J, Kudzia P, Long A, Hendron K, Holt KG, O'Donnell K, Ellis TD, Walsh CJ. Reducing Circumduction and Hip Hiking During Hemiparetic Walking Through Targeted Assistance of the Paretic Limb Using a Soft Robotic Exosuit. Am J Phys Med Rehabil. 2017 Oct;96(10 Suppl 1):S157-S164. doi: 10.1097/PHM.0000000000000800. PMID 28777105
- [Background] Awad LN, Bae J, O'Donnell K, De Rossi SMM, Hendron K, Sloot LH, Kudzia P, Allen S, Holt KG, Ellis TD, Walsh CJ. A soft robotic exosuit improves walking in patients after stroke. Sci Transl Med. 2017 Jul 26;9(400):eaai9084. doi: 10.1126/scitranslmed.aai9084. PMID 28747517
- [Background] Bae J, Awad LN, Long A, O'Donnell K, Hendron K, Holt KG, Ellis TD, Walsh CJ. Biomechanical mechanisms underlying exosuit-induced improvements in walking economy after stroke. J Exp Biol. 2018 Mar 7;221(Pt 5):jeb168815. doi: 10.1242/jeb.168815. PMID 29361587
- [Background] Ardestani MM, Kinnaird CR, Henderson CE, Hornby TG. Compensation or Recovery? Altered Kinetics and Neuromuscular Synergies Following High-Intensity Stepping Training Poststroke. Neurorehabil Neural Repair. 2019 Jan;33(1):47-58. doi: 10.1177/1545968318817825. Epub 2018 Dec 29. PMID 30595090
- [Background] Paci M. Physiotherapy based on the Bobath concept for adults with post-stroke hemiplegia: a review of effectiveness studies. J Rehabil Med. 2003 Jan;35(1):2-7. doi: 10.1080/16501970306106. PMID 12610841
- [Background] Roelker SA, Bowden MG, Kautz SA, Neptune RR. Paretic propulsion as a measure of walking performance and functional motor recovery post-stroke: A review. Gait Posture. 2019 Feb;68:6-14. doi: 10.1016/j.gaitpost.2018.10.027. Epub 2018 Oct 25. PMID 30408710
- [Background] Bowden MG, Balasubramanian CK, Neptune RR, Kautz SA. Anterior-posterior ground reaction forces as a measure of paretic leg contribution in hemiparetic walking. Stroke. 2006 Mar;37(3):872-6. doi: 10.1161/01.STR.0000204063.75779.8d. Epub 2006 Feb 2. PMID 16456121
- [Background] Bae J, Siviy C, Rouleau M, et al. A lightweight and efficient portable soft exosuit for paretic ankle assistance in walking after stroke. Proc - IEEE Int Conf Robot Autom. 2018:2820-2827. doi:10.1109/ICRA.2018.8461046
- [Background] Awad LN, Kudzia P, Revi DA, Ellis TD, Walsh CJ. Walking faster and farther with a soft robotic exosuit: Implications for post-stroke gait assistance and rehabilitation. IEEE Open J Eng Med Biol. 2020;1:108-115. doi: 10.1109/ojemb.2020.2984429. Epub 2020 Apr 2. PMID 33748765
- [Background] Porciuncula F, Arumukhom Revi D, Baker TC, et al. Speed-Based Gait Training with Soft Robotic Exosuits Improves Walking after Stroke: A Crossover Pilot Study. In: American Physical Therapy Association Combined Sections Meeting.; 2021.
- [Background] Kesar TM, Reisman DS, Higginson JS, Awad LN, Binder-Macleod SA. Changes in Post-Stroke Gait Biomechanics Induced by One Session of Gait Training. Phys Med Rehabil Int. 2015;2(10):1072. Epub 2015 Dec 28. PMID 27819067
- [Background] Awad LN, Reisman DS, Pohlig RT, Binder-Macleod SA. Identifying candidates for targeted gait rehabilitation after stroke: better prediction through biomechanics-informed characterization. J Neuroeng Rehabil. 2016 Sep 23;13(1):84. doi: 10.1186/s12984-016-0188-8. PMID 27663199
- [Background] Reisman D, Kesar T, Perumal R, Roos M, Rudolph K, Higginson J, Helm E, Binder-Macleod S. Time course of functional and biomechanical improvements during a gait training intervention in persons with chronic stroke. J Neurol Phys Ther. 2013 Dec;37(4):159-65. doi: 10.1097/NPT.0000000000000020. PMID 24189337
- [Background] Awad LN, Kesar TM, Reisman D, Binder-Macleod SA. Effects of repeated treadmill testing and electrical stimulation on post-stroke gait kinematics. Gait Posture. 2013 Jan;37(1):67-71. doi: 10.1016/j.gaitpost.2012.06.001. Epub 2012 Jul 15. PMID 22796242
- [Background] Sabut SK, Lenka PK, Kumar R, Mahadevappa M. Effect of functional electrical stimulation on the effort and walking speed, surface electromyography activity, and metabolic responses in stroke subjects. J Electromyogr Kinesiol. 2010 Dec;20(6):1170-7. doi: 10.1016/j.jelekin.2010.07.003. Epub 2010 Aug 6. PMID 20692180
- [Background] Koelewijn AD, Audu M, Del-Ama AJ, Colucci A, Font-Llagunes JM, Gogeascoechea A, Hnat SK, Makowski N, Moreno JC, Nandor M, Quinn R, Reichenbach M, Reyes RD, Sartori M, Soekadar S, Triolo RJ, Vermehren M, Wenger C, Yavuz US, Fey D, Beckerle P. Adaptation Strategies for Personalized Gait Neuroprosthetics. Front Neurorobot. 2021 Dec 16;15:750519. doi: 10.3389/fnbot.2021.750519. eCollection 2021. PMID 34975445
- [Background] Bajd T, Munih M. VI.2. Basic functional electrical stimulation (FES) of extremites - an engineer's view. Stud Health Technol Inform. 2010;152:343-52. PMID 20407203
- [Background] Embrey DG, Holtz SL, Alon G, Brandsma BA, McCoy SW. Functional electrical stimulation to dorsiflexors and plantar flexors during gait to improve walking in adults with chronic hemiplegia. Arch Phys Med Rehabil. 2010 May;91(5):687-96. doi: 10.1016/j.apmr.2009.12.024. PMID 20434604
- [Background] Kesar TM, Perumal R, Reisman DS, Jancosko A, Rudolph KS, Higginson JS, Binder-Macleod SA. Functional electrical stimulation of ankle plantarflexor and dorsiflexor muscles: effects on poststroke gait. Stroke. 2009 Dec;40(12):3821-7. doi: 10.1161/STROKEAHA.109.560375. Epub 2009 Oct 15. PMID 19834018
- [Background] Palmer JA, Hsiao H, Wright T, Binder-Macleod SA. Single Session of Functional Electrical Stimulation-Assisted Walking Produces Corticomotor Symmetry Changes Related to Changes in Poststroke Walking Mechanics. Phys Ther. 2017 May 1;97(5):550-560. doi: 10.1093/ptj/pzx008. PMID 28339828
- [Background] Awad LN, Reisman DS, Pohlig RT, Binder-Macleod SA. Reducing The Cost of Transport and Increasing Walking Distance After Stroke: A Randomized Controlled Trial on Fast Locomotor Training Combined With Functional Electrical Stimulation. Neurorehabil Neural Repair. 2016 Aug;30(7):661-70. doi: 10.1177/1545968315619696. Epub 2015 Nov 30. PMID 26621366
- [Background] Reisman DS, Binder-MacLeod S, Farquhar WB. Changes in metabolic cost of transport following locomotor training poststroke. Top Stroke Rehabil. 2013 Mar-Apr;20(2):161-70. doi: 10.1310/tsr2002-161. PMID 23611857
- [Background] Clark DJ, Ting LH, Zajac FE, Neptune RR, Kautz SA. Merging of healthy motor modules predicts reduced locomotor performance and muscle coordination complexity post-stroke. J Neurophysiol. 2010 Feb;103(2):844-57. doi: 10.1152/jn.00825.2009. Epub 2009 Dec 9. PMID 20007501
- [Background] Steele KM, Rozumalski A, Schwartz MH. Muscle synergies and complexity of neuromuscular control during gait in cerebral palsy. Dev Med Child Neurol. 2015 Dec;57(12):1176-82. doi: 10.1111/dmcn.12826. Epub 2015 Jun 17. PMID 26084733
- [Background] Collimore AN, Aiello AJ, Pohlig RT, Awad LN. The Dynamic Motor Control Index as a Marker of Age-Related Neuromuscular Impairment. Front Aging Neurosci. 2021 Jul 22;13:678525. doi: 10.3389/fnagi.2021.678525. eCollection 2021. PMID 34366824
- [Background] Collimore AN, Pohlig RT, Awad LN. Minimal viable muscle set for identifying impairments in the neuromuscular control of walking using the dynamic motor control index. In: North American Congress on Biomechanics. Ottawa, CA. 2022.
- [Background] Collimore AN, Aiello AJM, Pohlig RT, Awad LN. The dynamic motor control index is a better marker of age-related neuromotor impairments than the number of muscle synergies: Toward early detection of walking deficits. Neural Control of Movement Annual Meeting. Virtual. 2021.
- [Background] Choe DK, Aiello AJ, Spangler JE, Walsh CJ, Awad LN. A Propulsion Neuroprosthesis Improves Overground Walking in Community-Dwelling Individuals After Stroke. IEEE Open J Eng Med Biol. 2024 Jul 4;5:563-572. doi: 10.1109/OJEMB.2024.3416028. eCollection 2024. PMID 39157060